CLINICAL TRIAL: NCT06277804
Title: A Phase I Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LTC004 in Combination With Cyclophosphamide and Fludarabine in Patients With Advanced or Metastatic Malignancies Tumor
Brief Title: A Phase I Study of LTC004 Combin With FC in Patients With Advanced/Metastatic Malignancies Tumor
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Letolab (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LTC004-102
Record Dates: First submitted 2024-02-07; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Adult Solid Tumor
MeSH Terms: interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose-escalation phase (Experimental): LTC004 combined with fludarabine, cyclophosphamide, "3+3"design； LTC004 was given on day 1 and cyclophosphamide (250 mg/m2) combined with fludarabine (25 mg/m2) on days 3 and 4 of each cycle.Q3W.
  Interventions: Drug: LTC004 in Combination With Cyclophosphamide and Fludarabine
- Dose-expansion phase (Experimental): Further evaluation of the safety and efficacy of this dosing regimen in patients with sarcoma who have failed standard treatment according to the RP2D identified in Dose-escalation phase.
  Interventions: Drug: LTC004 in Combination With Cyclophosphamide and Fludarabine

INTERVENTIONS:
Drug: LTC004 in Combination With Cyclophosphamide and Fludarabine — LTC004 was given on day 1 and cyclophosphamide (250 mg/m2) in combination with fludarabine (25 mg/m2) was given on days 3 and 4 of each cycle, Q3W, until disease progression, withdrawn informed or intolerable

SUMMARY:
This was a multicenter, open PHASE I study of LTC004 in Combination With Cyclophosphamide and Fludarabine in Patients With Advanced/Metastatic Malignancies Tumor, the study design consisting of 2 phases: Phase Ia (Phase Ia dose escalation) and Phase Ib (Phase Ib expansion). The objective of this study was to evaluate combination safety, tolerability, pharmacokinetic,pharmacodynamics characteristics, and initial efficacy in advanced malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 75 years；
2. Subjects with a histologically or cytologically confirmed diagnosis of a locally advanced or metastatic solid tumor or lymphoma that is not amenable to surgical treatment at the time of screening and that has failed after standard treatment as recommended by existing clinical standards of care or guidelines or that is not refractory to standard treatment and/or for which there is no currently effective standard of care.

   The current open indication population is patients with soft tissue sarcoma, with the following specific requirements:

   Histologically/cytologically confirmed diagnosis of unresectable or metastatic soft tissue sarcoma with failure of existing standard therapy or lack of effective treatment, as follows: 1) For pathological subtypes other than adenovascular soft tissue sarcoma and epithelioid sarcoma, failure of, or intolerance to, at least standard chemotherapy regimens of adriamycin or adriamycin in combination with isocyclophosphamide; and 2) For adenovascular soft tissue sarcoma and epithelioid sarcoma. Prior treatment failure or intolerance to a targeted agent [anti-angiogenic class such as amlotinib, pezopanib, etc.] is required; Note: Disease progression <6 months after the end of treatment in neoadjuvant or adjuvant patients is considered first-line treatment;
3. At least one measurable tumor lesion based on RECIST V1.1 criteria；
4. ECOG PS ≤1；
5. Expected survival ≥12 weeks；
6. Adequate organ function；
7. Patients who have received any chemotherapy or anti-tumor monoclonal antibody drugs within 4 weeks prior to the first dose of study drug (excluding mitomycin and nitrosoureas within 6 weeks prior to the first dose of study drug）; small molecule targeted drugs within 2 weeks prior to the first dose of study drug; Chinese medicine therapy (Chinese medicine therapy with clear anti-tumor indications in the package insert ）within 4 weeks prior to the first dose of study drug；
8. Patients, both females and males, of reproductive potential must agree to use adequate contraception during and for 6 months after the last infusion of LTC004.
9. Understands and provides written informed consent and willing to follow the requirements specified in protocol.

Exclusion Criteria:

1. History of severe hypersensitivity reactions to other mAbs.
2. Untreated, unstable or uncontrolled central nervous system (CNS) metastases with following exceptions:A. Clinically stable MRI scans and no progressive or uncontrolled neurologic symptoms or signs for at least 4 weeks prior to the first study treatment;
3. Patients with uncontrolled pleural effusion, pericardial effusion or abdominal effusion as judged by the investigator at screening;
4. Patients with untreated or clinically symptomatic spinal cord compression that has not been controlled.
5. Previous immunotherapy, including IL-2, IL-15, PD-1/L1 inhibitors, NK, and TCR-T cell therapy；
6. ≥2 malignant tumors within 5 years prior to first dose of drug；
7. Moderate to severe dyspnea at rest, severe primary lung disease, current need for continuous oxygen therapy, or clinically active interstitial lung disease (ILD) or pneumonia due to advanced cancer or its complications; Grade ≥3 interstitial pneumonia during prior antineoplastic therapy；
8. Persons with active tuberculosis infection within 1 year prior to enrollment by history or screening, or persons with a history of active tuberculosis infection more than 1 year ago without regular treatment；
9. Presence of severe infection within 4 weeks prior to first dose of medication，Presence of active infection requiring systemic antibiotic therapy with CTCAE grade ≥2 within 2 weeks prior to first dose
10. History of serious cardiovascular disease；
11. Active hepatitis B (hepatitis B virus titer > lower limit of detection) or hepatitis C at the time of screening；
12. Syphilis-positive patients at screening；
13. Active, or previous autoimmune disease with potential for recurrence at the time of screening；
14. Immunodeficiency diseases or history of such diseases, including a positive serologic test for human immunodeficiency virus (HIV)；
15. Those who have experienced clinically significant bleeding symptoms within 3 months prior to the first dose of the drug；
16. Those who have received systemic immunosuppressive therapy (including but not limited to glucocorticoids, cyclophosphamide, azathioprine, methotrexate, thalidomide, etc.) within 2 weeks prior to the first dose;
17. Immunomodulatory medications within 2 weeks prior to first dose；
18. Those who received radical radiation therapy within 4 weeks prior to the first dose and those who received palliative radiation within 14 days prior to the first dose；
19. Tumor invasion into peripheral vital organs (e.g., aorta and trachea) or risk of esophageal-tracheal fistula or esophageal-pleural fistula; history of gastrointestinal perforation and/or fistula within 6 months prior to the first dose of the drug；
20. Received other unlisted clinical investigational drug or treatment within 4 weeks prior to first dose；
21. Use of live or attenuated vaccines within 4 weeks prior to the first dose, or anticipated need for live or attenuated vaccines during the study period；
22. Major surgery (other than surgery for diagnostic purposes) within 4 weeks prior to the first dose, anticipation of major surgery (other than surgery for diagnostic purposes) during the study period, or diagnostic or low-invasive surgery within 7 days prior to the first dose (excluded for puncture biopsies).
23. Adverse effects of prior antitumor therapy have not recovered to CTCAE version 5.0 grade rating ≤1；
24. Patients who have received a previous allogeneic bone marrow/hematopoietic stem cell transplant or solid organ transplant；
25. Pregnant and lactating women；
26. Subjects who in the judgment of the investigator, have a history of other serious systemic disease or are unfit to participate in this trial for any other reason (the presence of psychiatric disorders in the patient that may affect compliance with the trial, alcohol, drug or substance abuse, etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Safety, tolerability and antitumor efficacy of Combination. | up to 12 months
  Dose-limiting toxicity (DLT) Incidence;TEAE and SAE Incidence，Changes in safety indicators before and after administration

SECONDARY OUTCOMES:
PK Characteristics and immunogenicity of Combination | up to 12 months
  Serum concentration and antibody positivity of LTC004

IPD SHARING:
Plan to Share IPD: No